CLINICAL TRIAL: NCT04142840
Title: Comparing the Efficacy of Dexmedetomidine and Propofol in the Treatment of Emergence Agitation Occurring in Adults After General Anesthesia: A Randomised Control Trial DP-TEA Trial
Brief Title: Dexmedetomidine and Propofol in the Treatment of Emergence Agitation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DP-TEA Trial
Record Dates: First submitted 2019-10-19; First posted 2019-10-29 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-10

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Experimental): General anesthesia will be maintained by sevoflurane and remifentanil. End-tidal carbon dioxide will be controlled between 35 mmHg to 40 mmHg.Mean blood pressure(MAP) will be administrated between 80% and 120% of the baseline.Heart rate is going to be maintained between 50-100 beats per minute.
  In consultation with the surgeons and 5 minutes prior to the departure of the operating room,all the anesthesia agents are discontinued and the patient will be transferred to the post-anaesthesia care unit.And reversal agents are given to antagonize the residual muscular relaxant.Once emergence agitation occurs,the patient assigned to the dexmedetomidine group will be infused with a single dose of 0.7ug/kg dexmedetomidine.
  Interventions: Drug: Dexmedetomidine
- Propofol Group (Active Comparator): General anesthesia will be maintained by sevoflurane and remifentanil. End-tidal carbon dioxide will be controlled between 35 mmHg to 40 mmHg.Mean blood pressure(MAP) will be administrated between 80% and 120% of the baseline.Heart rate is going to be maintained between 50-100 beats per minute.
  In consultation with the surgeons and 5 minutes prior to the departure of the operating room,all the anesthesia agents are discontinued and the patient will be transferred to the post-anaesthesia care unit.And reversal agents are given to antagonize the residual muscular relaxant.Once emergence agitation occurs,the patient assigned to the propofol group will be infused with a single dose of 0.5mg/kg propofol.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — a selective α-2 adrenoceptor agonist which is widely used as an adjuvant to general anesthesia
  Arms: Dexmedetomidine Group
Drug: Propofol — a short -acting medication that result in a decreased level of consciousness and lack of memory for events,widely used including the starting and maintenance of general anesthesia.
  Arms: Propofol Group

SUMMARY:
1. This clinical research aims to compare the effects of dexmedetomidine and propofol on the treatment of emergence agitation in adult patients after general anesthesia.
2. Half of participants will receive dexmedetomidine while the other half will receive propofol when emergence agitation happens.

DETAILED DESCRIPTION:
As a common problem observed in pediatric patients after sevoflurane anesthesia, emergence agitations are investigated mainly in children.For adults,previous studies were almost about the efficacy of premedication on preventing emergence agitation. Once emergence agitation happens, there is still no guidelines established to recommend the medication usage in the post-anaesthesia care unit.So high-quality prospective clinical studies are required to provide evidence for emergence agitation treatment.

Dexmedetomidine and propofol are both widely used in general anesthesia and can be acquired easily.When emergence agitation occurs,both injections are common choices in daily clinical administration on emergence agitation.To the investigator's knowledge ,propofol with a very quick onset is superior for anesthesia goals, but is without analgesia effects.While dexmedetomidine can produce sedation,analgesia,anxiolysis.So the investigators propose the hypothesis here that dexmedetomidine is prior to propofol on the treatment of emergence agitation in adults patients after general anesthesia.Therefore this research is undertaken to verify the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 years old after general anesthesia
* with informed consent provided.

Exclusion Criteria:

* age younger than 18 years or older than 65 years;
* American Society of Anesthesiologists classification ≥Ⅲ;
* preoperative lung dysfunction(including pneumonia,atelectasis,adult respiratory distress syndrome,acute lung injury and so on);
* preoperative heart dysfunction(including sever cardiac coronary disease,unstable angina,LVEF≤30％，sick sinus syndrome，bradycardia:heart rate≤50bpm,second or third degree A-V block);
* history of mental disease;
* no informed consent provided;
* uncontrolled hypertension(baseline blood pressure:SBP≥160mmHg or DBP≥110mmHg);
* cancers;
* enrolled in other researches within 90 days;
* allergic to intervening medicine.
* BMI less than 18 or more than 30 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate of emergence agitation assessed by the Riker Sedation-Agitation Scale after the treatment of each group. | 1 day
  1. The Riker Sedation-Agitation Scale is raging from a maximum value of 7 to a minimum value of 1.Lower scores mean a better outcome.
  2. A Riker Sedation-Agitation scale score of 5 or more than 5 will be considered as emergence agitation.

SECONDARY OUTCOMES:
Riker Sedation-Agitation Scale scores before and after intervention; | 1 day
  Riker Sedation-Agitation Scale is raging from a maximum value of 7 to a minimum value of 1.Lower scores mean a better outcome.
Heart rate before and after intervention; | 1 day
  Heart rate wil be recorded in beats per minute.
The consumption of sufentanil in the post-anaesthesia care unit; | 1 day
  During the procedure,a dose of 0.01ug/kg sulfentanil will be given when numeric rating scale scores≥ 5 scores or the patient has a analgesia request; Numeric rating scale,with a maximum value of 10 and a minimum value of 0,is specifically as follows:0-3,slight pain;4-7,moderate pain;8-10,sever pain.Lower scores mean a better outcome.
Nausea and vomiting scores when leaving the post-anesthesia care unit. | 1 day
  According the following scale with a maximum value of 3 and a minimum value of 0,is specifically as follows:0,no nausea;1,mild nausea;2,sever nausea requiring antiemetics;3,retching,vomiting or both.Lower scores mean a better outcome.
Duration in the post-anaesthesia care unit | 1 day
  The total time from entering the post-anaesthesia care unit to leaving the post-anaesthesia care unit.
Recovering quality: recovery scale | 24 hours after surgery.
  The recovering quality is evaluated by the 40-item quality of recovery scale,with a maximum value of 200 and a minimum value of 0.Higher scores mean a better outcome.
Mean blood pressure before and after intervention; | 1 day
  Mean blood pressure will be recorded in millimeters of mercury.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital,Shanghai Jiao Tong University,School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Feng Z, Shi X, Yan X, Zhu Y, Gu J, Zhu H, Yu W, Zhang S. Comparing the effects of dexmedetomidine versus propofol on the treatment of emergence agitation in adult patients after general anesthesia: study protocol for a randomized, superiority, controlled trial (DP-TEA Trial). Trials. 2021 Nov 16;22(1):811. doi: 10.1186/s13063-021-05743-2. PMID 34784941